CLINICAL TRIAL: NCT05066425
Title: Soluble Corn Fiber for Promoting Executive Function Study
Acronym: SCOPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Tate and Lyle Ingredients Americas LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 21839
Record Dates: First submitted 2021-07-27; First posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-07

CONDITIONS: Health
Keywords: Microbiota; Cognition; Fiber
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Soluble Corn Fiber (Experimental): 22g Soluble Corn Fiber/day for 4 weeks
  Interventions: Dietary Supplement: Soluble Corn Fiber
- Maltodextrin (Placebo Comparator): 22g Maltodextrin/day for 4 weeks
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Soluble Corn Fiber — Participants will be asked to consume a packet of 22g Soluble Corn Fiber/day for 4 weeks
  Arms: Soluble Corn Fiber
Dietary Supplement: Maltodextrin — Participants will be asked to consume a packet of 22g Maltodextrin/day for 4 weeks
  Arms: Maltodextrin

SUMMARY:
The overarching aim of this study is to test the influence of daily consumption of a soluble corn fiber (SCF) known i.e., PROMITOR® Soluble Fibre™ for cognitive function among middle and older-aged adults.

DETAILED DESCRIPTION:
Although regular consumption of soluble dietary fiber has been shown to support multiple markers of gastrointestinal and physical health, the effects of regular fiber consumption for promoting cognitive health remain unclear. Additionally, the GI microbiota-dependent mechanisms by which dietary fiber may impact markers of cognitive function remain understudied. Thus, the overarching aim of this study is to test the influence of daily consumption of a soluble corn fiber (SCF) known i.e., PROMITOR® Soluble Fibre™ for cognitive function among middle and older-aged adults. The primary hypothesis is that daily consumption of dietary fiber over a period of 4 weeks will significantly improve executive function. The secondary hypothesis is that the influence of SCF on cognitive outcomes will be mediated by improvement in GI bacterial taxa and fermentation-end product profiles. These hypotheses will be tested by conducting a 4 week randomized, double-blind, placebo-controlled cross-over study among healthy, i.e., free-living cognitively intact middle-aged and older adults between45-75 years of age. This work is significant because most Americans do not meet their recommended dietary fiber intake and there is a growing interest in understanding the potential benefits of consuming dietary fiber for broader health outcomes including both gastrointestinal and cognitive health.

ELIGIBILITY:
Inclusion Criteria:

1. 45-75 years of age
2. Free of cognitive impairment (Mini-Mental State Examination score of higher than 24)
3. Absence of neurological disease
4. Absence of gastrointestinal diseases
5. Absence of prediabetes or diabetes
6. No color blindness
7. Have normal or corrected-to-normal vision
8. No history of antibiotics or smoking over the past 3 months
9. Agree to refrain from taking pre-or probiotic supplements during the study
10. Agree to inform researchers of any changes in chronic medications during the study
11. Body Mass Index (BMI) between 18.5 to 34.9 kg/m2
12. Habitual dietary fiber consumption of ≤12g/d (women) and ≤19 g/d (men) based on DHQ II
13. Not consuming an extreme dietary pattern (e.g., vegan, keto, low FODMAP)
14. No allergies to corn or maltodextrin, eggs, peanuts, tree nuts, wheat and soy
15. Agree to maintain habitual dietary patterns throughout the study period
16. Maintain their current level of physical activity
17. Complete all necessary study questionnaires and to provide stool specimens as required.

Exclusion Criteria:

1. <45 or >75 years of age
2. Presence of cognitive impairment (Mini-Mental State Examination score of lower than 24)
3. Presence of neurological disease
4. Presence of gastrointestinal diseases
5. Presence of prediabetes or diabetes
6. Color blindness
7. Non normal or uncorrected vision
8. History of antibiotics or smoking over the past 3 months
9. Not agree to refrain from taking pre- or probiotic supplements during the study
10. Not agree to communicate any changes in chronic medications during the study
11. Body Mass Index (BMI) below 18.5 or greater than 34.9 kg/m2
12. Habitual dietary fiber consumption of >12g/d (women) and >19 g/d (men) based on DHQ II
13. Consuming an extreme dietary pattern (e.g., vegan, keto, low FODMAP)
14. Allergies to corn and/or maltodextrin
15. Not agree to maintain habitual dietary patterns throughout the study period
16. Not agree to maintain their current level of physical activity
17. Not agree to complete all necessary study questionnaires and to provide stool specimens as required.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-08-02 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Attention Accuracy | 4 weeks
  Behavioral performance measured as accuracy (%) during Flanker task
Attention Reaction Time | 4 weeks
  Behavioral performance measured as response time (ms) during Flanker task
P3 Amplitude | 4 weeks
  Amplitude (microvolt) of the P3 ERP waveform assessed during the Flanker task
Event-related potentials | 4 weeks
  Latency (ms) of the P3 ERP waveform assessed during the Flanker task
Relational Memory | 4 weeks
  Accuracy during a spatial reconstruction task

SECONDARY OUTCOMES:
Gastrointestinal Microbiota | 4 weeks
  Taxonomic compositionprofiles of the gastrointestinal microbiota
Fecal Metabolites | 4 weeks
  Quantity of short-chain fatty acids in fecal samples
Mood/Well-being | 4 weeks
  Total score on surveys (POMS, PANAS, SF-36)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No